CLINICAL TRIAL: NCT05243550
Title: A Phase 3, Single-Arm, Multicenter Study to Evaluate the Efficacy and Safety of UGN-102 as Primary Chemoablative Therapy in Patients With Low-Grade (LG) Non-Muscle Invasive Bladder Cancer (NMIBC) at Intermediate Risk (IR) of Recurrence
Brief Title: A Phase 3 Single-Arm Study of UGN-102 for Treatment of Low-Grade Intermediate-Risk Non-Muscle Invasive Bladder Cancer
Acronym: ENVISION
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL011
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Bladder Cancer; Urothelial Carcinoma; Urothelial Carcinoma Bladder
Keywords: Non-muscle invasive bladder cancer; Low grade non-muscle invasive bladder cancer; Intermediate risk non-muscle invasive bladder cancer; NMIBC; UGN-102; Mitomycin
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Non-Muscle Invasive Bladder Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UGN-102 (Experimental): Patients will receive 6 once-weekly intravesical instillations of UGN-102 (75 mg mitomycin).
  Interventions: Drug: UGN-102

INTERVENTIONS:
Drug: UGN-102 — UGN-102 consists of mitomycin and sterile hydrogel (a proprietary thermally responsive gel) that is used to reconstitute mitomycin before instillation. The reverse thermal properties of UGN-102 allow for local administration of mitomycin as a liquid under chilled conditions, with subsequent conversion to a semi-solid gel depot following instillation into the bladder.
  Other Names: UGN-102 (mitomycin) for intravesical solution

SUMMARY:
This Phase 3, multinational, single-arm study was designed to evaluate the efficacy and safety of UGN-102 as primary chemoablative therapy in patients with recurrent low-grade intermediate-risk non-muscle invasive bladder cancer (LG-IR-NMIBC).

DETAILED DESCRIPTION:
Eligible patients received 6 once-weekly intravesical instillations of UGN-102.

All patients returned to the clinic approximately 3 months after the first instillation for determination of response to treatment. Assessment of response was based on visual observation (white light cystoscopy), histopathology of any remaining or new lesions by central pathology lab (if applicable), and interpretation of urine cytology by central pathology lab.

Patients who had a complete response (CR) at the 3-month Visit, defined as having no detectable disease in the bladder, entered the Follow-up Period of the study. Patients who had a non-complete response (NCR) due to residual LG disease underwent investigator-designated standard of care (SOC) treatment of remaining lesions and then entered the Follow-up Period of the study.

During the Follow-up Period, patients return to the clinic every 3 months for up to 24 months (ie, 27 months after the first instillation) for evaluation of response. Patients who remain disease free at the 27-month Visit will continue to be followed every 6 months for up to 36 months (ie, 63 months after the first instillation) or until disease recurrence, disease progression, death, or the study is closed by the sponsor, whichever occurs first.

Patients who had a disease recurrence during the Follow-up Period or a disease progression at any time underwent investigator-designated SOC treatment and had a separate End of Study (EOS) Visit performed. The timing of the EOS Visit was approximately 3 months after SOC treatment of disease recurrence or progression.

Study conduct is ongoing and data are summarized through a cutoff date of 04 Apr 2024. As of the data cutoff date, ongoing patients were followed through at least Study Month 15, with the earliest enrolled patients followed through Study Month 21.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and the protocol.
2. Patient who has LG-NMIBC (Ta) histologically confirmed by cold cup biopsy at Screening or within 8 weeks before Screening.
3. History of LG-NMIBC requiring treatment with transurethral resection of bladder tumors (TURBT). Note: This refers to a previous episode(s) and not to the current episode for which the patient is being screened.
4. Has intermediate-risk disease, defined as having 1 or 2 of the following:

   * Presence of multiple tumors;
   * Solitary tumor > 3 cm;
   * Early or frequent recurrence (≥ 1 occurrence of LG-NMIBC within 1 year of the current diagnosis at the initial Screening Visit).
5. Negative voiding cytology for high-grade (HG) disease within 8 weeks before Screening.
6. Has adequate organ and bone marrow function as determined by routine laboratory tests as below:

   * Leukocytes ≥ 3,000 per μL;
   * Absolute neutrophil count ≥ 1,500 per μL;
   * Platelets ≥ 100,000 per μL;
   * Hemoglobin ≥ 9.0 g/dL;
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN);
   * Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 × ULN;
   * Alkaline phosphatase ≤ 2.5 × ULN;
   * Estimated glomerular filtration rate ≥ 30 mL/min.
7. Has an anticipated life expectancy of at least the duration of the trial.
8. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Women of childbearing potential (defined as premenopausal women who have not been sterilized), including female patients and female partners of male patients, must be willing to use 2 acceptable forms of effective contraception from enrollment through 6 months post-treatment.

Exclusion Criteria:

1. Received Bacillus Calmette-Guérin treatment for urothelial carcinoma (UC) within previous 1 year.
2. History of HG bladder cancer (papillary or carcinoma in situ) in the past 2 years.
3. Known allergy or sensitivity to mitomycin that in the Investigator's opinion cannot be readily managed.
4. Clinically significant urethral stricture that would preclude passage of a urethral catheter.
5. History of:

   * Neurogenic bladder;
   * Active urinary retention;
   * Any other condition that would prohibit normal voiding.
6. Past or current muscle invasive bladder cancer (ie, T2, T3, T4) or metastatic UC.
7. Current tumor grading of T1.
8. Concurrent upper tract UC.
9. Evidence of active urinary tract infection that in the Investigator's opinion cannot be treated and resolved prior to biopsy and/or administration of study treatment.
10. Is pregnant or breastfeeding.
11. Has an underlying substance abuse or psychiatric disorder such that, in the opinion of the Investigator, the patient would be unable to comply with the protocol.
12. History of prior treatment with an intravesical chemotherapeutic agent in the past 2 years except for a single dose of chemotherapy immediately after any previous TURBT.
13. Has participated in a study with an investigational agent or device within 30 days of enrollment.
14. Has previously participated in a study in which they received UGN-102.
15. Has any other active malignancy requiring treatment with systemic anticancer therapy (eg, chemotherapy, immunotherapy, radiation therapy). Superficial cancers such as cutaneous basal cell or squamous cell carcinomas that can be treated locally are allowed.
16. Has any other clinically significant medical or surgical condition that in the Investigator's opinion could compromise patient safety or the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2028-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sandip Prasad, MD, Principal Investigator — Atlantic Health System
Locations (65):
- United States (16):
  - Arizona Urology Specialists, Tucson, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - Genesis Research, San Diego, California
  - Wichita Urology Group, Wichita, Kansas
  - John Hopkins University, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - University of Missouri, Columbia, Missouri
  - Atlantic Health System, Morristown, New Jersey
  - Great Lakes Physician dba WNY Urology Associates, Cheektowaga, New York
  - AccuMed Research Associates, Garden City, New York
  - Manhattan Medical Research, New York, New York
  - NYU Langone Health, New York, New York
  - Mount Sinai, New York, New York
  - Urology Associates, P.C., Nashville, Tennessee
  - Houston Methodist Research Institute, Houston, Texas
  - Spokane Urology, P.S., Spokane, Washington
- Medical University Vienna, Department of Urology, Vienna, Austria
- Bulgaria (18):
  - Multiprofile Hospital for Active Treatment - Blagoevgrad, Blagoevgrad
  - Multiprofile Hospital for Active Treatment "Dr. Tota Venkova", Gabrovo, Department of Urology, Gabrovo
  - Multiprofile Hospital for Active Treatment "Sveti Nikolai Chudotvorets", Lom, Lom
  - Multiprofile Hospital for Active Treatment "City Clinic - Sveti Georgi", Montana
  - University Multiprofile Hospital for Active Treatment "Dr. Georgi Stranski", Pleven, Urology Clinic, Pleven
  - University Multiprofile Hospital for Active Treatment "Sveta Marina" - Pleven, Department of Urology, Pleven
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv, Plovdiv
  - University Multiprofile Hospital for Active Treatment, Plovdiv, Plovdiv
  - Multiprofile Hospital for Active Treatment Park Hospital, Plovdiv
  - University Multiprofile Hospital for Active Treatment 'Kanev', Ruse, Department of Urology, Rousse
  - Multiprofile Hospital for Active Treatment - Shumen, Shumen, Department of Urology, Shumen
  - University Multiprofile Hospital for Active Treatment "Tsaritsa Yoanna - ISUL", Sofia, Sofia
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine "N.I. Pirogov", Sofia, Urology Clinic, Sofia
  - Multiprofile Hospital for Active Treatment - Targovishte, Targovishte
  - Multiprofile Hospital for Active Treatment "Life Hospital" Burgas, Varna
  - Multiprofile Hospital for Active Treatment, Varna part of Military Medical Academy, Clinic of Urology, Varna
  - Multiprofile Hospital for Active Treatment "Sveta Anna", Varna, Urology Clinic, Varna
  - Multiprofile Hospital for Active Treatment "Sveti Pantaleymon", Yambol, Department of Urology, Yambol
- Estonia (5):
  - East Viru Central Hospital, Surgery Clinic, Kohtla-Järve
  - East Tallinn Central Hospital Ltd., Surgery Clinic, Centre of Urology, Tallinn
  - West Tallinn Central Hospital Ltd., Department of Urology, Tallinn
  - North Estonia Medical Centre Foundation Ltd., Surgery Clinic, General and Oncology Urology Centre, Tallinn
  - Tartu University Hospital, Surgery Clinic, Department of Urology and Kidney Transplantation, Tartu
- Georgia (5):
  - LTD Central University Clinic After Academic N. Kipshidze, Tbilisi
  - JSC Jerarsi, Department of Urology, Tbilisi
  - LTD Gidmedi, Urology Department, Tbilisi
  - Pineo Medical Ecosystem Ltd., Department of Urology, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Technology Medical Center University Clinic LTD, Urology Department, Tbilisi
- Latvia (4):
  - Liepajas Regional Hospital, Urology Department, Liepāja
  - P. Stradins Clinical University Hospital, Center for Urology, Riga
  - LLC Riga East University Hospital, Clinic of Urology and Oncologic Urology, Riga
  - Daugavpils Regional Hospital, Urology Department, Riga
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas
  - Klaipeda University Hospital, Klaipėda
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Poland (4):
  - AKMED, Gliwice
  - SCM sp. z o.o. (LLC), Krakow
  - Clinical Research Center Limited liability company Medic-R Limited partnership, Poznan
  - Mazovian Oncology Hospital, Subdepartment of Urology, Wieliszew
- Serbia (4):
  - Clinical Center of Serbia, Clinic of Urology, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Clinic of Surgery, Department of Urology, Belgrade
  - Clinical Hospital Center Zemun, Urology unit, Belgrade
  - Clinical Center Kragujevac, Clinic of Urology, Nephrology and Dialysis, Kragujevac
- Spain (5):
  - Hospital del Mar, Barcelona
  - Hospital de Basurto, Bilbao
  - University Hospital Foundation Jimenez Diaz, Madrid
  - University Hospital 12 de Octubre, Madrid
  - La Paz University Hospital, Madrid

REFERENCES:
- [Result] Prasad SM, Shishkov D, Mihaylov NV, Khuskivadze A, Genov P, Terzi V, Kates M, Huang WC, Louie MJ, Raju S, Burger B, Meads A, Schoenberg M. Primary Chemoablation of Recurrent Low-Grade Intermediate-Risk Nonmuscle-Invasive Bladder Cancer With UGN-102: A Single-Arm, Open-Label, Phase 3 Trial (ENVISION). J Urol. 2025 Feb;213(2):205-216. doi: 10.1097/JU.0000000000004296. Epub 2024 Oct 24. PMID 39446087
- [Derived] Stover AM, Mueller D, Carda-Auten J, Hilton A, Tsurutis V, Smith AB. Perceived Impact on Patient Routines/Responsibilities for Surgery and a Nonsurgical Primary Treatment Option in Recurrent Low-Grade Intermediate-Risk Nonmuscle-Invasive Bladder Cancer: Findings From the ENVISION Phase 3 Trial. J Urol. 2025 Jul;214(1):18-31. doi: 10.1097/JU.0000000000004511. Epub 2025 Mar 6. PMID 40048558

RESULTS

PARTICIPANT FLOW:
Groups:
- UGN-102: 6 once-weekly intravesical instillations of UGN-102 (75 mg mitomycin).
Period: Overall Study
Arm/Group | UGN-102
Started | 240
Completed | 43
Not Completed | 197
Not completed — Ongoing in the Study | 171
Not completed — Withdrawal by Subject | 10
Not completed — Lost to Follow-up | 7
Not completed — Adverse Event | 3
Not completed — Noncompliance | 1
Not completed — Physician Decision | 1
Not completed — Other Reason | 4

BASELINE CHARACTERISTICS:
Population: All patients who received any dose of UGN-102.
Arm/Group | UGN-102
Number analyzed (Participants) | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 78
  >=65 years | 162
Age, Continuous [Median (Full Range); unit: years] | 70 [30 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 147
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 237
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 234
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Bulgaria | 85
  United States | 41
  Latvia | 38
  Georgia | 20
  Serbia | 18
  Estonia | 14
  Spain | 8
  Lithuania | 7
  Poland | 7
  Austria | 2
Previous Low-grade Non-muscle Invasive Bladder Cancer (LG-NMIBC) Episode(s) [Count of Participants; unit: Participants]
  Yes | 229
  No | 11
Previous LG-NMIBC Episode(s) Within 1 Year [Count of Participants; unit: Participants]
  Yes | 124
  No | 116
Prior Transurethral Resection of Bladder Tumor (TURBT) to Treat LG-NMIBC [Count of Participants; unit: Participants]
  Yes | 228
  No | 12
Longest Tumor Diameter [Count of Participants; unit: Participants] — Longest tumor diameter is defined as the longest diameter among all measurable lesions.
  Participants
    ≤ 3 cm | 216
    > 3 cm | 19
    Missing | 5
Tumor Burden [Count of Participants; unit: Participants] — Tumor burden is defined as the sum of the longest diameters of measurable lesions.
  Participants
    ≤ 3 cm | 180
    > 3 cm | 41
    Missing | 19
Tumor Count [Count of Participants; unit: Participants]
  Single | 41
  Multiple | 198
  Missing | 1
Smoking History [Count of Participants; unit: Participants] — Smoker category includes both former and current smokers. Non-smoker category includes "Never."
  Participants
    Non-smoker | 112
    Smoker | 128

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as the percentage of patients who achieved a complete response (CR) at the 3-month Visit. A patient was considered a CR if there was no detectable disease in the bladder based on visual observation (white light cystoscopy), biopsy of remaining lesions (if applicable), and voiding urine cytology.
Time Frame: 3 months
Population: All patients who received any dose of UGN-102.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UGN-102
Number analyzed (Participants) | 240
percentage of participants | 76.7 [70.8 to 81.9]

2. Secondary Outcome: Duration of Response (DOR) in Patients Who Achieved CR at the 3-month Visit
Description: DOR is defined as the time from the first documented CR to the earliest date of recurrence or progression as determined using the date of cystoscopy, for cause biopsy, or cytology, or death due to any cause, whichever occurred first.
Time Frame: Up to 60 months
Reporting Status: Not Posted

3. Secondary Outcome: Durable Complete Response (DCR) Rate in Patients Who Achieved CR at the 3-month Visit
Description: DCR rate at scheduled disease assessment time points is defined as the percentage of patients who had a CR at the 3-month Visit and maintained CR up to that particular follow-up visit.
Time Frame: Up to 60 months
Reporting Status: Not Posted

4. Secondary Outcome: Disease-free Survival (DFS) in Patients Who Achieved CR at the 3-month Visit
Description: DFS is defined as the time from the first instillation to the earliest date of recurrence or progression as determined using the date of cystoscopy, for cause biopsy, or cytology, or death due to any cause, whichever occurred first.
Time Frame: Up to 63 months
Reporting Status: Not Posted

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs of Special Interest
Description: The number of patients with each type of event is summarized. TEAEs were defined as adverse events (AEs) that started on or after the day of the first instillation of UGN-102 or pre-treatment AEs that worsened during the study.
Time Frame: Up to 21 months
Population: All patients who received any dose of UGN-102.
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102
Number analyzed (Participants) | 240
Participants
  Any TEAEs | 137
  Any serious TEAEs | 29
  Any TEAEs of special interest | 100

6. Secondary Outcome: Number of Participants With Post-baseline Potentially Clinically Significant (PCS) Hematology Values
Description: The number of patients with each type of event is summarized.
Time Frame: 6 months
Population: All patients who received any dose of UGN-102 and who had a post-baseline laboratory value, except for hemoglobin, which required non-missing laboratory values at baseline and post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102
Number analyzed (Participants) | 240
Participants
  Hemoglobin < 0.8 × lower limit of normal and > 20% decrease from baseline: number analyzed (Participants) | 238
  Hemoglobin < 0.8 × lower limit of normal and > 20% decrease from baseline | 8
  Hemoglobin > 1.3 × upper limit of normal (ULN) and > 30% increase from baseline: number analyzed (Participants) | 238
  Hemoglobin > 1.3 × upper limit of normal (ULN) and > 30% increase from baseline | 0
  Lymphocytes < 0.5 × 10^9/L | 1
  Lymphocytes > 20 × 10^9/L | 0
  Neutrophils < 1.0 × 10^9/L | 1
  Platelets < 75 × 10^9/L | 1
  Platelets ≥ 700 × 10^9/L | 0
  Leukocytes ≤ 2.8 × 10^9/L | 2
  Leukocytes ≥ 16.0 × 10^9/L | 5

7. Secondary Outcome: Number of Participants With Post-baseline PCS Chemistry Values
Description: The number of patients with each type of event is summarized.
Time Frame: 6 months
Population: All patients who received any dose of UGN-102 and who had a post-baseline laboratory value.
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102
Number analyzed (Participants) | 240
Participants
  Alanine aminotransferase > 3 × ULN | 1
  Aspartate aminotransferase > 3 × ULN | 1
  Bilirubin > 1.5 × ULN | 6
  Creatinine > 194 μmol/L | 8
  Gamma glutamyl transferase > 2.5 × ULN | 11
  Potassium < 3.0 mmol/L | 0
  Potassium > 5.5 mmol/L | 20
  Sodium ≤ 130 mmol/L | 1
  Sodium > 150 mmol/L | 0

ADVERSE EVENTS:
Time Frame: Up to 21 months. Study conduct is ongoing and data are summarized through a cutoff date of 04 Apr 2024. As of the data cutoff date, ongoing patients were followed through at least Study Month 15, with the earliest enrolled patients followed through Study Month 21.
Description: Adverse events (AEs) were reported from the time of informed consent to the 6-month Visit. After the 6-month Visit, all serious AEs (regardless of causality) and non-serious AEs assessed as related to study treatment or study procedures were to be reported until the End of Study Visit.
Arm/Group | UGN-102
All-Cause Mortality (participants affected / at risk) | 3/240
Serious Adverse Events (participants affected / at risk) | 29/240
Other Adverse Events (participants affected / at risk) | 129/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UGN-102 (N=240)
Atrial fibrillation (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Atrioventricular block second degree (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
COVID-19 (Infections and infestations) | 2
Fournier's gangrene (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Carotid artery disease (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urinary retention (Renal and urinary disorders) | 2
Urethral stenosis (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Gallbladder polyp (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Glaucoma (Eye disorders) | 1
Death (General disorders) | 1
Blood creatinine increased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UGN-102 (N=240)
Dysuria (Renal and urinary disorders) | 54
Haematuria (Renal and urinary disorders) | 20
Pollakiuria (Renal and urinary disorders) | 16
Urinary retention (Renal and urinary disorders) | 11
Urinary tract infection (Infections and infestations) | 17
Fatigue (General disorders) | 13
Urethral stenosis (Renal and urinary disorders) | 11
Micturition urgency (Renal and urinary disorders) | 8
Constipation (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT05243550/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT05243550/SAP_001.pdf